CLINICAL TRIAL: NCT03263546
Title: Implementation of Internet-delivered Cognitive-behavior Therapy for Paediatric Obsessive-compulsive Disorder in the Clinic: a Randomized Stepped Care Non-inferiority Trial
Brief Title: Internet-delivered CBT for Paediatric OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Eva Serlachius, MD, associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REPN 2017/1070-31/1
Record Dates: First submitted 2017-08-18; First posted 2017-08-28 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stepped care (Experimental): Internet-delivered cognitive behavioral therapy (ICBT)
  Interventions: Behavioral: Internet-delivered cognitive behavioral therapy (ICBT)
- Gold standard treatment (Active Comparator): Cognitive behavioral therapy (CBT)
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Internet-delivered cognitive behavioral therapy (ICBT) — Participants will receive internet-delivered CBT with therapist support for 16 weeks. The treatment consists of 14 online chapters with interactive features as videos and illustrations. The treatment has the main focus on exposure with ritual prevention. The children and parents have regular contact with a personal assigned therapist via written text messages in the platform.
  Participants that are classified as non-responders at 3 months follow-up will receive face-to-face CBT of up to 12 sessions over 12 weeks.
  Arms: Stepped care
Behavioral: Cognitive behavioral therapy (CBT) — Participants in the gold standard group will receive 14 individual face-to-face CBT sessions over 16 weeks. The treatment is based on current evidence based recommendations for OCD, and focuses on exposure with ritual prevention.
  Participants that are classified as non-responders at 3 months follow-up will receive additional face-to-face CBT of up to 12 sessions over 12 weeks.
  Arms: Gold standard treatment

SUMMARY:
The purpose of this study is to investigate if therapist-guided internet-delivered cognitive behavioral therapy (ICBT) in a stepped-care approach is an effective and cost-effective treatment in reducing OCD symptoms for children and adolescents compared to gold standard treatment (face-to-face CBT).

DETAILED DESCRIPTION:
A randomized controlled non-inferiority trial comparing therapist-guided internet-delivered cognitive behavioral therapy (ICBT) in a stepped care model with face-to-face CBT for children and adolescents with obsessive-compulsive disorder (OCD).

Participants will be randomized to either stepped care ICBT or to gold standard face-to-face CBT. One group (stepped care) will be first offered ICBT for 16 weeks. Non-responders at the 3-month follow-up will receive additional face-to-face CBT. The other group (gold standard treatment) will be randomized directly to receive face-to-face CBT for 16 weeks. Non-responders will, as in the other group, receive additional face-to-face treatment after the 3-month follow-up. The primary endpoint will be at 6-month follow-up. Long-term effects are also investigated (1 year, 2 years and 5 years after treatment completion).

The primary objective is to evaluate whether ICBT in a stepped care approach will be non-inferior to gold standard treatment (face-to-face CBT) in reducing OCD symptoms, depression, impairment, sleep problems, health and functioning. The secondary objective is to a) carry out a full health economic evaluation and b) investigate if self-referred and referred participants differ regarding outcome in the two treatment groups.

The hypotheses are:

1. An ICBT stepped care approach will be non-inferior to gold standard treatment (face-to-face CBT) in reducing OCD symptoms.
2. The stepped care approach will be associated with lower costs, such as reduced therapist and administration times, service utilization, minimized work and school absence for families etc., compared to gold standard treatment.
3. Self-referred patients will benefit significantly better than referred patients regarding outcome in the ICBT group, but there will not be any difference in the face-to-face CBT group.

ELIGIBILITY:
Inclusion Criteria:

* Primary DSM-5 diagnosis of OCD
* Total score of ≥16 on the Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS)
* Age between 7 and 17 years
* Ability to read and write Swedish and with access to a computer and use of internet.
* Participants on psychotropic medication must had been on a stable dose for the last 6 weeks prior to baseline assessment. If the child is on medication for OCD, they will be requested to stay on stable doses for the duration of the trial.

Exclusion Criteria:

* Organic brain disorders, global learning disabilities, autism spectrum disorder, psychosis, bipolar disorder and severe eating disorder.
* Suicidal ideation
* Not able to understand the basics of the ICBT self-help material, patient being housebound or in need of intensive- or in-patient treatment.
* Having completed a course of CBT for OCD within the last 12 months (defined as at least 5 sessions CBT including exposure and response prevention).
* Children with ongoing psychological treatment for OCD or another anxiety disorder will not be included in the study.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Children's Yale Brown Obsessive-Compulsive Scale (CY-BOCS) | week 0, week 16, at 3 and 6 months follow-up, at 1, 2 and 5 years follow-up.
  Change in OCD symptom severity from baseline to week 16 and 3 and 6 months after treatment has ended, and at 1, 2 and 5 years follow-up. Primary endpoint is 6 months follow-up.

SECONDARY OUTCOMES:
Clinical global impression severity (CGI-S) | week 0, week 16, at 3 and 6 months follow-up, at 1, 2 and 5 years follow-up
  Change in global severity from baseline to week 16 and 3 and 6 months after treatment has ended, and at 1, 2 and 5 years follow-up.
Clinical global impression improvement (CGI-I) | week 16, at 3 and 6 months follow-up, at 1, 2 and 5 years follow-up
  Change in global improvement from week 16 to 3 and 6 months after treatment has ended, and at 1, 2 and 5 years follow-up.
Children's global assessment scale (C-GAS) | week 0, week 16, at 3 and 6 months follow-up, at 1 year follow-up
  Change in global functioning from baseline to week 16 and 3 and 6 months after treatment has ended, and at 1 year follow-up.
Obsessive-compulsive inventory - child version (OCI-CV) | week 0, week 16, at 3 and 6 months follow-up, at 1 year follow-up, and weekly during treatment
  Change in child-rated OCD symptoms from baseline to week 16 and 3 and 6 months after treatment has ended, at 1 year follow-up, and weekly during treatment.
The Child Health Utility 9D (CHU9D) | week 0, week 16, at 3 and 6 months follow-up, at 1 year follow-up
  Change in general health from baseline to week 16 and 3 and 6 months after treatment has ended, and at 1 year follow-up.
Insomnia Severity Index (ISI) | week 0, week 16, at 3 and 6 months follow-up, at 1 year follow-up
  Change in sleep problems from baseline to week 16 and 3 and 6 months after treatment has ended, and at 1 year follow-up
Children's Obsessional Compulsive Inventory Revised - parent version (ChOCI-R) | week 0, week 16, at 3 and 6 months follow-up, at 1 year follow-up, and weekly during treatment
  Change in parent-rated OCD symptoms from baseline to week 16 and 3 and 6 months after treatment has ended, at 1 year follow-up, and weekly during treatment.
Family accommodation scale for obsessive-compulsive disorder - self-rated version (FAS-SR) | week 0, week 16, at 3 and 6 months follow-up, at 1 year follow-up
  Change in parent-rated family accommodation from baseline to week 16 and 3 and 6 months after treatment has ended, and at 1 year follow-up
Trimbos/iMTA questionnaire for Costs associated with Psychiatric Illness (TiC-P) | week 0, week 16, at 3 and 6 months follow-up, at 1, 2 and 5 years follow-up.
  Change in economic costs from baseline to week 16 and 3 and 6 months after treatment has ended, and at 1, 2 and 5 years follow-up.
Mood and Feeling Questionnaire (MFQ) | week 0, week 16, at 3 and 6 months follow-up, at 1 year follow-up
  Change in child and parent rated depressive symptoms from baseline to week 16 and 3 and 6 months after treatment has ended, and at 1 year follow-up
Education, work and social adjustment scale (EWSAS) | week 0, week 16, at 3 and 6 months follow-up, at 1 year follow-up
  Change in child and parent rated impairment and functioning from baseline to week 16 and 3 and 6 months after treatment has ended, and at 1 year follow-up

OTHER OUTCOMES:
Autism Spectrum Quotient (AQ-10) | week 0
  Measure of autistic symptoms at baseline
Treatment credibility and expectancy scale | week 2
  Child and parent version. Investigate if both conditions have equal credibility in order to rule out placebo.
Working alliance inventory (WAI) | week 2
  Child and parent version. Investigate if both conditions have equal working alliance in order to rule out non-specific factors.
Client Satisfaction Questionnaire (CSQ-8) | week 16 and at 6 months follow-up
  Child and parent version. Investigate if both conditions have equal satisfaction.
Patient EX/RP Adherence Scale (PEAS) | week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12, week 13, week 14, week 15, week 16
  Clinician-rated version during face-to-face CBT. Self-rated version during both ICBT and face-to-face CBT. Investigate treatment adherence in both conditions.
internet intervention Patient Adherence Scale (iiPAS) | week 8 and 16
  Investigate treatment adherence in the ICBT condition.
Parental strategy scale | week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12, week 13, week 14, week 15, week 16
  Investigate the use of parental strategies weekly during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Serlachius, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - BUP Specialmottagning, Gothenburg
  - Child and Adolescent Psychiatry (CAP) research center, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aspvall K, Andersson E, Melin K, Norlin L, Eriksson V, Vigerland S, Jolstedt M, Silverberg-Morse M, Wallin L, Sampaio F, Feldman I, Bottai M, Lenhard F, Mataix-Cols D, Serlachius E. Effect of an Internet-Delivered Stepped-Care Program vs In-Person Cognitive Behavioral Therapy on Obsessive-Compulsive Disorder Symptoms in Children and Adolescents: A Randomized Clinical Trial. JAMA. 2021 May 11;325(18):1863-1873. doi: 10.1001/jama.2021.3839. PMID 33974020
- [Derived] Aspvall K, Andersson E, Lenhard F, Melin K, Norlin L, Wallin L, Silverberg-Morse M, Feldman I, Bottai M, Mataix-Cols D, Serlachius E. Stepped Care Internet-Delivered vs Face-to-Face Cognitive-Behavior Therapy for Pediatric Obsessive-Compulsive Disorder: A Trial Protocol for a Randomized Noninferiority Trial. JAMA Netw Open. 2019 Oct 2;2(10):e1913810. doi: 10.1001/jamanetworkopen.2019.13810. PMID 31642928